CLINICAL TRIAL: NCT06725095
Title: Effects of Enamel Matrix Derivative in the Non-surgical Mechanical Debridement Treatment of Peri-implant Mucositis
Brief Title: Effects of Enamel Matrix Derivative in the Treatment of Peri-implant Mucositis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-3306
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Mucositis; Peri Implant Mucositis
Keywords: Enamel matrix derivative
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator: non-surgical sub-marginal peri-implant instrumentation (NSPI) with placebo gel (Placebo Comparator): Patients received a one-session of non-surgical sub-marginal peri-implant instrumentation (NSPI) with placebo
  Interventions: Other: Placebo gel
- non-surgical sub-marginal peri-implant instrumentation (NSPI) with EMD (Active Comparator): Patients received a one-session of non-surgical sub-marginal peri-implant instrumentation (NSPI) with EMD
  Interventions: Other: Enamel Matrix Proteins Derivative

INTERVENTIONS:
Other: Placebo gel — Patients were treated with non surgical peri-implant mucositis therapy with non-surgical sub-marginal peri-implant instrumentation plus the use of a placebo gel
  Arms: Placebo Comparator: non-surgical sub-marginal peri-implant instrumentation (NSPI) with placebo gel
Other: Enamel Matrix Proteins Derivative — Patients were treated with non surgical peri-implant mucositis therapy with non-surgical sub-marginal peri-implant instrumentation plus the use of non-surgical treatment plus Enamel Matrix Proteins Derivative
  Arms: non-surgical sub-marginal peri-implant instrumentation (NSPI) with EMD

SUMMARY:
To evaluate the naturally occurring peri-implant mucositis (PM) treatment by means of non-surgical sub-marginal peri-implant instrumentation (NSPI) with or without use of enamel matrix protein derivative (EMD). Specifically, the primary outcome of the present study compared the efficacy of NSPI +EMD with respect to NSPI and placebo in the treatment of PM at 6 months follow-up by means of BOP reduction. The secondary outcome evaluated the influence of possible predictors on the BOP changes among all follow-up sessions.

DETAILED DESCRIPTION:
Patients (n° 54) with Implants affected by PM were randomly assigned to test (NSMD+EMD) or control procedures (NSMD + placebo). At baseline, 1, 3, 6 months, full-mouth plaque score (FMPS), full-mouth bleeding score (FMBS), probing depth (PD), bleeding on probing (BOP), modified gingival index (mGI), and modified plaque index (mPlI) will assessed as well as levels of periodontal bacteria such as Aggregatibacter Actynomycencomitans, Porphyromonas Gingivalis, Tannerella Forsythia and Treponema Denticola. The BOP reduction was set as a primary outcome and the patient was considered statistical unit. Data were analysed to assess BOP reduction at a 6-month follow-up and to identify significant predictors of implant-site BOP through mixed generalized linear regression.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old;
* implants with smooth necks supporting cemented or screw-retained single-unit crowns with at least one BOP-positive site (Berglundh et al., 2018),
* implants placed in both maxilla and mandible
* patients with gingivitis or treated periodontitis with the absence of residual PD ≥5 mm
* presence at least of 2 mm of keratinized mucosa (KT) at implant sites

Exclusion Criteria:

* presence of systemic diseases;
* pregnancy or lactating;
* use of inflammatory drugs or antibiotics within 3 months prior to study recruitment;
* implants with modified (i.e., micro-rough) necks;
* interproximal open contacts between implant restoration and adjacent teeth; peri-implantitis (Berglundh et al., 2018)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) changes | 6-months
  The number of implants presenting with complete absence of BOP or implants with limited extent of BOP (≤1 spot/implant-the presence of a single spot)

SECONDARY OUTCOMES:
Probing pocket depth (PPD) changes | 6-months
  Changes in PPD
Full mouth plaque score (FMPS) % changes | 6-months
  Full mouth plaque score (FMPS) % changes
Full mouth bleeding score (FMBS) % changes | 6-months
  Changes in FMBS
Plaque at implant sites according to modified gingival index (mGI) changes score | 6-months
  Changes in mGI 0-4 score
Plaque at implant sites according to modified plaque index (mPlI) changes score | 6-months
  Changes in mPlI 0-4 score
Patient-Reported Outcome Measures (PROMs) | 6-months
  Patient-Reported Outcome Measures (PROMs) Were evaluated PROMs such as the number of abscesses, systemic complications, gingival recession, excessive bleeding, allergic effects, systemic impacts and related drug side effects

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, DDS, Principal Investigator — University of Catania
Locations (1):
- Policlinico G. Rodolico, Catania, Ct, Italy

IPD SHARING:
Plan to Share IPD: Yes
Pubmed
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: pubmed databse
URL: https://pubmed.ncbi.nlm.nih.gov/